CLINICAL TRIAL: NCT06376149
Title: A Pilot Randomized-controlled Trial Evaluating the Efficacy of a Live-Online Mindfulness-Based Intervention: The Making Mindfulness Matter© in Children With Juvenile Idiopathic Arthritis Study
Brief Title: M3-JIA: Making Mindfulness Matter for Children With JIA
Acronym: M3-JIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Brain Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 124973
Record Dates: First submitted 2024-04-03; First posted 2024-04-19 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-03

CONDITIONS: Juvenile Idiopathic Arthritis; Children; Mental Health; Mental Well-being
Keywords: M3; mindfulness
MeSH Terms: conditions — Arthritis, Juvenile; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The primary objective is to conduct a pilot RCT to evaluate the effectiveness of a live-online mindfulness-based family intervention program, Making Mindfulness Matter (M3©) for children with JIA and their caregiver(s).
  Measures will be obtained via questionnaires at 3 time points for the intervention group: baseline, 9 weeks and 2 months post-intervention. For the control group questionnaires will be obtained 4 time points: baseline, 9 weeks, 18 weeks and 2 months post intervention.
  Additionally, at the start of each session, parents will complete a one-page semi-structured questionnaire evaluating treatment fidelity and at home utilization of M3© skills. At the end of each session, parent participants will complete a one-page structured questionnaire providing feedback on the session, and facilitators will complete the M3© Adherence Checklist, evaluating whether planned activities were completed, and any modifications made.
Who Masked: Participant, Care Provider
Masking Description: Participants will be blinded to their group assignment: all participants will be told that they will receive the intervention. Program facilitators will be blinded to participant group assignment order, since sessions for both study arms would run on a rolling basis. The statistician will also be blinded to the group assignment and order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Intervention Group (Other): Child-parent dyads will undergo a standardized 8-week course of Making Mindfulness Matter© (M3). The program will be delivered online using live, interactive sessions to groups of 4 to 8, for 1.5 hours each week for the parent group and 1 hour each week for the child group. Children and parents will attend separate on-line sessions and at the end of each child session, the parent will be asked to join their child on-line for a shared mindful exercise. Once 4 to 8 dyads are assigned to the intervention group, participants will be given the baseline questionnaires and start the intervention in the following week.
  Interventions:
  Behavioural: Making Mindfulness Matter© (M3)
  Interventions: Behavioral: M3 Intervention group
- Other: Waitlist Control (Other): Child-parent dyads randomized to the control arm will continue treatment as usual. Once 4 to 8 dyads are assigned to the control group, participants will be given the baseline questionnaires, They will complete Follow-up questionnaire and extended follow up questionnaires at comparable times to families in the intervention arm. With one extra set of questionnaires at the completion of the intervention. These dyads will be provided with the intervention at the next scheduled session; the goal is to provide the intervention to controls as soon as possible to avoid differential attrition between the intervention and control arm. During the intervention sessions, they will complete all feasibility surveys pertaining to the intervention and their satisfaction with each intervention session.
  Interventions:
  Behavioural: Making Mindfulness Matter© (M3)
  Interventions: Behavioral: M3 Waitlist Group

INTERVENTIONS:
Behavioral: M3 Intervention group — The M3© program offered online concurrently for parents and children (4-12 years of age). Each parent session is 90 minutes long, and each child session is 60 minutes long. Parents and children learn similar concepts, at developmentally appropriate levels.
  Arms: Experimental: Intervention Group
Behavioral: M3 Waitlist Group — The M3© program offered online concurrently for parents and children (4-12 years of age). Each parent session is 90 minutes long, and each child session is 60 minutes long. Parents and children learn similar concepts, at developmentally appropriate levels.
  Arms: Other: Waitlist Control

SUMMARY:
The investigator will evaluate the efficacy of M3©, an intervention for patients with JIA and their caregivers. Children with Juvenile arthritis and their parents will attend an 8 week online program called Making Mindfulness Matter (M3). This is a facilitator-led program that integrates knowledge and skills related to mindfulness, social-emotional learning, neuroscience, and positive psychology to promote coping and resiliency for children and families in context of the challenges of pediatric chronic disease. The child program is designed for children 4-12 years of age, with each lesson including a variety of concrete ways to teach children skills based on their age/developmental level.

DETAILED DESCRIPTION:
This pilot RCT is essential to refine the implementation of the intervention to families with a child with JIA and collect information pertaining to the feasibility and effectiveness of the intervention in preparation for a subsequent multicentred trial across Canada. The investigator will propose to test if the M3© program improves the child's health related quality of life (HRQOL) and mental health for Children with JIA and caregivers. Additionally, to address the knowledge gap on the relationship between mental health and disease outcomes in JIA. M3 is a promising mindfulness-based intervention which may have mental health benefits for children with JIA and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 12 years diagnosed with JIA
* Children have reasonable comprehension of spoken language and can follow simple instructions
* Children with JIA and their caregivers are willing to attend intervention sessions and have access to technology and internet to attend the online sessions.
* Children with JIA and their caregivers have an adequate understanding of English

Exclusion Criteria:

* Other major co-morbid disorders (e.g. Crohn's disease, diabetes, renal failure).
* Concurrent enrollment in other intervention trials or practicing any complementary health interventions such as yoga, meditation, or daily mindfulness practice.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
conduct a pilot RCT to evaluate the effectiveness of a live-online mindfulness-based family intervention program, Making Mindfulness Matter (M3©) for children with JIA and their caregiver(s). | Throughout the study enrollment period and over the 8 weeks of intervention.
  At the start of each session, parents will complete a one-page (12-item) semi-structured questionnaire evaluating treatment fidelity, at home utilization of M3 skills. At the end of each session, parents will complete an overall feedback form on the intervention. Facilitators will complete a two-page questionnaire providing feedback on the session. At the start and end of the M3 program, children will be asked to complete a feeling face questionnaire rated on a 3-point scale about topics discussed in the group such as how our brain works when upset and what is mindfulness. The minimum score being 0 with the highest score being 10 where the higher the score means the better the outcome.

SECONDARY OUTCOMES:
Effects of M3 on health related quality of life of children with JIA | baseline, 9 weeks, 18 weeks and 2 months later.
  Peds Quality of life (PedsQL) is a 23-item measure for children ages 2-18 years that emphasizes a functional approach to quality of life by examining the child's sense of well-being and ability to engage in physical and social activities, to concentrate, think and remember, and to regulate behaviour. Generates an overall Peds-QL score, and four subscale scores: cognitive, emotional, social, and physical functioning. Parent report is obtained for children <6 years old.
  The investigators will calculate the minimum clinically important difference (MCID). To calculate the MCID for the Peds-QL, the Patient Centred Global Ratings of Change will be used, a 5-item scale where respondents indicate the amount of change relative to baseline. Rating from -7 (much worse) through 0 (no change) to +7 (much better). This information will allow us to calculate the MCID for the Ped-QL, and thereby identify the proportion of patients who experience a clinically meaningful change following intervention.
Effects of M3 on health quality of life for parents | baseline, 9 weeks, 18 weeks and 2 months later.
  The Peds-QL Family Impact module is a 36-item measure designed to measure the impact of pediatric chronic health conditions on parents and the family. It measures parent self-reported physical, emotional, social, and cognitive functioning, communication, and worry, as well as parent-reported family daily activities and family relationships. Generates an overall score. Items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better outcomes.
Does M3 have a positive effect on children's severity of JIA | baseline, 9 weeks, 18 weeks and 2 months later.
  The pediatric Symptom check list is a 17-question screening tool that is used to improve the recognition and treatment of psycho social problems in children ages 4 to 17 years as a parent reported measure.
  The total score is calculated by adding together the score for each of the 17 items. A score of 15 and over is considered at risk.
Does M3 have a positive effect on children's executive function | baseline, 9 weeks, 18 weeks and 2 months later.
  Behavioral Rating Inventory of Executive Function 2 (BRIEF) 63-item scale measuring parent-rated executive function and self-regulation in children. Generates a global executive composite, cognitive regulation index, emotion regulation index, behavior regulation index. Persons with T-score above 60 in a given scale are categorized as 'at-risk' for that domain.

OTHER OUTCOMES:
Does M3 have a positive effect on parents' stress | baseline, 9 weeks, 18 weeks and 2 months later.
  Parenting Stress Index 4 - short form 36-item scale that helps identify sources of stress. Focused on three major domains of stress: child characteristics, parent characteristics, and situational/demographic factors. A summary and 3 subscale (Parental Distress, Parent-Child Dysfunctional Interaction and Difficult Child) scores are generated. Scores in the 81st percentile or higher are indicative of high stress.
Does M3 have a positive effect on parents' depression and anxiety | baseline, 9 weeks, 18 weeks and 2 months later.
  The PROMIS- short forms- depression, anxiety is an 8 question measures for parents personal physical, mental, and social well-being.
  Each item on the measure is rated on a 5-point scale with a range in score from 7 to 35 with higher scores indicating greater severity of depression and anxiety.
Does M3 have a positive effect on Child's' depression and anxiety | baseline, 9 weeks, 18 weeks and 2 months later.
  The Revised Child Anxiety and Depression scale- (RCADS) is a 47-item, youth self-report (ages 8-18 years) questionnaire with subscales including: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and major depressive disorder. Parent report is obtained for children <8 years old.
  Scores below 65 are in the clinically normal range. Scores between 66-69 are in the boardline clinical range and scores above 70 are in the clinical range.
Does M3 have a positive effect on children's resiliency | baseline, 9 weeks, 18 weeks and 2 months later.
  Child &Youth Resiliency Measure (CYRM-R) is a 28 item resiliency self-report measure (ages 5-23 years). It looks at social ecological resiliency in children and adults.
  The possible range of scores for the total measure is 17 to 85, with higher scores indicating greater resilience.
Does M3 have a positive effect on parent resiliency | baseline, 9 weeks, 18 weeks and 2 months later.
  Connor Davidson-resilience scale (CD-RISC) is a 25 item measure that looks at resilience or how well one is equipped to bounce back after stressful events, tragedy, or trauma.
  evaluated on a five-point Likert scale ranging from 0 to 4: these ratings result in a number between 0-100, and higher scores indicate higher resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Berard, MD, Principal Investigator — LHSC Children's Hospital/ Lawson Research
Locations (3):
- Canada (3):
  - McMaster Children's Hospital,, Hamilton, Ontario
  - LHSC Children' Hosptial, London, Ontario
  - Sickids, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schonert-Reichl KA, Oberle E, Lawlor MS, Abbott D, Thomson K, Oberlander TF, Diamond A. Enhancing cognitive and social-emotional development through a simple-to-administer mindfulness-based school program for elementary school children: a randomized controlled trial. Dev Psychol. 2015 Jan;51(1):52-66. doi: 10.1037/a0038454. PMID 25546595
- [Background] Puka K, Bax K, Andrade A, Devries-Rizzo M, Gangam H, Levin S, Nouri MN, Prasad AN, Secco M, Zou G, Speechley KN. A live-online mindfulness-based intervention for children living with epilepsy and their families: protocol for a randomized controlled trial of Making Mindfulness Matter(c). Trials. 2020 Nov 11;21(1):922. doi: 10.1186/s13063-020-04792-3. PMID 33176853
- [Background] Treemarcki EB, Danguecan AN, Cunningham NR, Knight AM. Mental Health in Pediatric Rheumatology: An Opportunity to Improve Outcomes. Rheum Dis Clin North Am. 2022 Feb;48(1):67-90. doi: 10.1016/j.rdc.2021.09.012. PMID 34798960